CLINICAL TRIAL: NCT06336252
Title: Technology Assisted Nudging to Increase Physical Activity Among Hospitalised Medical Patients in Hospital and 3 Months After Discharge
Brief Title: Technology Assisted Nudging to Increase Physical Activity Among Hospitalised Medical Patients
Acronym: SENS4ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: AAL (Unknown); Innovationsfonden (Unknown)
Responsible Party: Principal Investigator, Christian Dall, Associate professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F-23059441
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: COPD; Heart Failure; Parkinson Disease; Arthritis; Old Age; Cachexia; Stroke Sequelae
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Parkinson Disease; Arthritis; Cachexia

STUDY DESIGN:
Intervention Model Description: 1/1 allocation
Who Masked: Outcomes Assessor
Masking Description: Primary outcome (accelerometer data) blinded for the investigator and assesor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 digital nudging (Experimental): In hospital Participants in the intervention group will receive usual hospital care and be provided with a sensor collecting data on physical activity level during hospitalisation AND a monitor placed at their bedside that displays information about their physical activity level, in terms of time spent bedridden, sitting, standing, and walking. This information will be visible to the health personnel, the patients, and their relatives. This feedback system is developed and provided by SENS Innovation.
  After discharge The visual feedback system from SENS will be continued after discharge and include an E-sport biking system provided by 4Mvideo. This integrated new system will combine an ergometer bike or sofa bike installed in the patient's own home or nursing home, and data from the sensor that the participants continue to wear after discharge will go into the SENS system, feeding back a visual track of their activities
  Interventions: Behavioral: Digital nudging intervention target to change behavior
- Arm 2 usual care (No Intervention): The participants in the non-exposed cohort will receive usual hospital care and be provided with a sensor collecting data on activity level during hospitalisation.

INTERVENTIONS:
Behavioral: Digital nudging intervention target to change behavior — In hospital Participants in the intervention group will receive usual hospital care and be provided with a sensor collecting data on physical activity level during hospitalisation AND a monitor placed at their bedside that displays information about their physical activity level, in terms of time spent bedridden, sitting, standing, and walking. This information will be visible to the health personnel, the patients, and their relatives. This feedback system is developed and provided by SENS Innovation.
  After discharge The visual feedback system from SENS will be continued after discharge and include an E-sport biking system provided by 4Mvideo. This integrated new system will combine an ergometer bike or sofa bike installed in the patient's own home or nursing home, and data from the sensor that the participants continue to wear after discharge will go into the SENS system, feeding back a visual track of their activities
  Arms: Arm 1 digital nudging

SUMMARY:
Primary Objective To investigate if patients hospitalised for older adults with a decreased level of physical function, either related to a chronic condition e.g., COPD, Congestive heart failure, renal failure; infections; frailty and tendency of falling; orthopaedic surgery - after hip fracture will increase their time spent out of bed during hospitalisation and 3 months after discharge through visual feedback and motivational intervention about physical activities from a new mobile technology.

Hypothesis Patients hospitalised for medical disease will increase their physical activity level during hospitalisation and 3 months after discharge through visual feedback and motivational intervention from a new mobile technology.

DETAILED DESCRIPTION:
STUDY DESIGN Description of the protocol The study will be conducted as a randomised multicentre trial including 3 hospitals in Europe (Copenhagen, Stavanger, and Genova). Patients admitted to Department of Respiratory Medicine, Department of Cardiology, and Department of Geriatrics, Department of Orthopaedic disease or Department of Neurology will be included, and they will have their physical activity level measured either with or without a monitor providing visual feedback of time spent bedridden, sitting, standing, and walking. After discharge the feedback will include an ergometer bike or sofa bike connected to the feedback mechanism.

Design A randomised multicentre study design is chosen. All participants will have their physical activity measured during hospitalisation and after discharge. Approximately half of the participants will receive visual feedback about the amount of physical activity from a mobile device placed on the bedside table while hospitalized, and after discharge, they will be provided with an ergometer bike or sofa bike connected to the feedback mechanism.

Allocation of participants The allocation of participants will be done 1 to 1, stratified by age group, gender, and level of mobility, to the control group (no feedback) and intervention group (visual feedback group). We schedule, that 162 patients will be possible to include in the analysis set (54 patients are planned to be included in Denmark, Norway, and Italy). A computer-generated randomisation sequence will be used to assign the participants in each site to the intervention and control arms.

Duration of study participation Each participant will be observed from admission of hospitalisation or until he/she is discharged and followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

An individual will be eligible for study participation if he/she meets the following criteria:

Aged ≥60

1. Is admitted to one of the participating departments
2. Has signed informed consent
3. Reads and speaks Danish, Norwegian, Italian, or English

Exclusion Criteria:

An individual will be excluded from the study if he/she meets any of the following criteria:

1. Any condition that, in the opinion of the investigator, makes the person unfit for participation, e.g., delirium and/or psychotic symptoms; moderate or severe depression (GDS>8 (short form)); major surgery; moderate/severe dementia (MoCA≤18); chemotherapy or radiation treatment ongoing at enrolment; moderate/severe frailty (CFS≥6)
2. Expected hospitalisation less than 24 hours
3. Has allergy towards band aid
4. Enrolled in any other clinical study within the duration of the current study.

While these criteria represent the criteria for being observed, only patients observed for at least 24 hours are included in the analysis population. For practical reasons it is not possible to predict those patients eligible for the analysis population at inclusion. Hence, we will monitor more patients than we will analyse (see statistical analysis section).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Time spent out of bed measured in minutes related to the total accelerometer wear time (minutes) | 3 month
  To assess physical activity a small tri-axial accelerometers is used. The accelerometer measures activity data in minutes per day.

SECONDARY OUTCOMES:
Readmission within 90 days | 3 month
  Number of readmissions 90 days following discharge
Length of stay (days) | 3 month assessment
  Days of hospitalization
Time spent lying down, sitting, standing, and walking measured in minutes related to the total accelerometer wear time (minutes) | 3 month
  Measured by objective accelerometer
Time spent out of bed in hospital in minutes related to the total accelerometer wear time (minutes) | 3 month assessment
  Measured by objective accelerometer
Time spent out of bed after discharge in minutes related to the total accelerometer wear time (minutes) | 3 month
  Measured by objective accelerometer
Quality of life (EQ5D-5L) | 3 month
  PROM quality of life, increase means better quality of life score
- In-hospital fall incidents | 3 month assessment
  Number of falls

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Christian Dall, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to Danish legislation